CLINICAL TRIAL: NCT05978557
Title: A Feasibility Study to Determine if a Novel Patient-derived Explant Platform Can Produce Drug Sensitivity Scores Within a Clinically Relevant Time Frame in Patients With CNS Tumors
Brief Title: Brain Slice Explants to Predict Drug Response in Brain Tumors
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2212
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Central Nervous System Tumor
Keywords: patient-derived explant; tissue
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biospecimen collection — Biospecimen will be collected during surgery.

SUMMARY:
This biospecimen collection study will evaluate the feasibility of engrafting and testing resected Central nervous system (CNS) tumors tumor tissue ex vivo to estimate drug response, in pediatric and adult subjects. CNS tumors display remarkable heterogeneity and unfortunately there are no reliable precision oncology platforms that can identify the most effective therapy for each patient. Recent work has demonstrated the success of functional precision oncology platforms using patient-derived explant (PDE) at predicting drug response in various cancers. Since PDEs maintain important aspects of tumor heterogeneity they may prove effective as functional models for CNS tumors. The purpose of this study is to explore the feasibility of using a novel PDE platform to generate drug sensitivity scores from patients with central nervous system tumors in Pediatric and adult subjects having low- or high-grade CNS tumors resected. The secondary objective is to estimate the proportion of successfully scaled PDEs generated per given tumor size.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

1. Written informed consent obtained to participate in the study and HIPAA authorization for the release of personal health information or written assent and parental consent for pediatric subjects or surrogate consent provided by the subject's legally authorized guardians.
2. A diagnosis of a tumor residing in the central nervous system with surgery plan to have surgical resection.
3. The subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designer.

Exclusion Criteria:

1. All subjects must not meet any of the following exclusion criteria prior to enrollment to participate in this study:

   Any serious medical or psychiatric disorder that would interfere with the subject's ability to give informed consent.
2. Incarcerated individuals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult subjects having low- or high-grade central nervous system tumors resected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of specimens yielding scores | Up to 28 days
  The proportion of evaluable specimens yielding patient-derived explant (PDE) drug sensitivity scores. Specimens will be collected during surgery for tumor resection. Excised specimens will be processed to generate PDE-based functional drug screening models. A panel of therapeutics will be chosen for each specimen according to pre-set criteria determined.

SECONDARY OUTCOMES:
The scalability of evaluable specimens | Up to 28 days
  The percentage of evaluable specimens amenable to proportionally scaled patient-derived explant (PDE) generation per specimen size will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Satterlee, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials